CLINICAL TRIAL: NCT00423735
Title: Phase II Trial of Dasatinib in Patients With Recurrent Glioblastoma Multiforme
Brief Title: Dasatinib in Treating Patients With Recurrent Glioblastoma Multiforme or Gliosarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: Radiation Therapy Oncology Group (Network); NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00744; NCI-2009-00744 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000526070; RTOG 0627 (Other: NRG Oncology); RTOG-0627 (Other: CTEP); U10CA180868 (NIH); U10CA021661 (NIH)
Record Dates: First submitted 2007-01-16; First posted 2007-01-18 (Estimated); Results first posted 2015-01-06 (Estimated); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Adult Giant Cell Glioblastoma; Adult Glioblastoma; Adult Gliosarcoma; Recurrent Adult Brain Neoplasm
MeSH Terms: conditions — Glioblastoma; Gliosarcoma; Brain Neoplasms | interventions — Dasatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (dasatinib) (Experimental): Patients receive dasatinib PO BID on days 1-28. Courses repeat every 28 days in the absence of disease progression and unacceptable toxicity.
  Interventions: Drug: Dasatinib; Other: Pharmacological Study

INTERVENTIONS:
Drug: Dasatinib — Given PO
  Other Names: BMS-354825; Sprycel
Other: Pharmacological Study — Correlative studies

SUMMARY:
This phase II trial studies how well dasatinib works in treating patients with glioblastoma multiforme or gliosarcoma that has come back. Dasatinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the therapeutic efficacy of dasatinib in all patients (i.e., stages 1B and 2 combined) with recurrent/progressive glioblastoma (GBM) as measured by 6-month progression-free survival.

SECONDARY OBJECTIVES:

I. To determine the therapeutic efficacy of dasatinib for stage 1B patients with recurrent/progressive GBM as measured by a hybrid endpoint of 6-month progression-free survival OR objective response of (complete response [CR] or partial response [PR]) rate.

II. To determine patient overall survival. III. To determine the toxicity of dasatinib in the treatment of patients with GBM.

IV. To determine radiographic response rate to treatment. V. To determine patient progression-free survival. VI. To explore molecular correlates of clinical outcome. VII. To explore pharmacokinetic correlates of dosing, toxicity, and efficacy.

OUTLINE:

Patients receive dasatinib orally (PO) twice daily (BID) on days 1-28. Courses repeat every 28 days in the absence of disease progression and unacceptable toxicity.

After the completion of study treatment, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven diagnosis of GBM; gliosarcoma is also an eligible diagnosis
* The patient must consent to submission of tissue for central pathology review
* Patients who have already undergone central pathology review through their enrollment on another Radiation Therapy Oncology Group (RTOG) GBM trial do not need to consent to having their material re-reviewed by the central pathologist for this study
* All patients must consent to molecular analysis of pre-dasatinib tumor tissue
* Patients accrued to stage I (closed to accrual) or stage IB (opened to accrual May 5, 2009) must have tumors overexpressing at least 2 known dasatinib targets (i.e., SRC proto-oncogene, non-receptor tyrosine kinase [SRC], v-kit Hardy-Zuckerman 4 feline sarcoma viral oncogene homolog [KIT], platelet-derived growth factor receptor [PDGFR], or ephrin type-A receptor 2 [EPHA2])
* Patients accrued to stage II (cohort closed; not currently applicable) do not require overexpression of SRC, KIT, PDGFR, or EPHA2
* History and physical examination, including height and weight, within 10 days prior to registration on study
* Brain magnetic resonance imaging (MRI) with and without gadolinium within 10 days prior to registration on study
* Contrast-enhanced computed tomography (CT) scans are allowed for patients who cannot undergo MRI scanning
* Karnofsky performance status >= 60
* Absolute neutrophil count (ANC) >= 1,000 cells/mm^3
* Platelets >= 75,000 cells/mm^3
* Hemoglobin (Hgb) >= 8.0 g/dl; (note: the use of transfusion or other intervention to achieve Hgb >= 8.0 g/dl is acceptable)
* Leukocytes >= 3,000 cells/mm^3
* Absolute lymphocyte count (ALC) >= 500 cells/mm^3
* Total bilirubin =< 1.5 X institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 institutional upper limit of normal
* Creatinine =< 3 X institutional upper limit of normal or creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* All patients must have undergone prior treatment with radiotherapy and temozolomide; no other prior treatments are allowed
* There must be unequivocal radiographic evidence for tumor progression by MRI or CT scan, and the same type of scan (i.e., MRI or CT) must be used throughout the period of protocol treatment for tumor measurement; patients must be on a stable or decreasing dose of corticosteroids for at least 5 days before the baseline MRI/CT is performed
* Patients having undergone recent surgery for recurrent/progressive disease are eligible as long as they have recovered from the effects of surgery; patients who recently underwent resection without measurable disease post-operatively are also eligible
* Measurable disease is not required for eligibility in patients who recently underwent resection as long as the following conditions are met as applicable:

  * Progression of disease led to the surgery
  * Gliadel wafers were not placed during the most recent surgery
  * Neither convection enhanced delivery nor catheters for infusion of chemotherapy were used during the most recent surgery
  * Radioactive seeds were not placed during the most recent surgery
  * The histology of the most recent surgery documented recurrent/persistent/progressive malignant glioma
* Women of childbearing potential must have a negative beta human chorionic gonadotropin (B HCG) pregnancy test =< 3 days prior to registration
* Patient must sign study-specific informed consent prior to study entry

Exclusion Criteria:

* Prior invasive malignancy (except non-melanomatous skin cancer) unless disease free for a minimum of 3 years; (for example, carcinoma in situ of the breast, oral cavity, or cervix are all permissible)
* Radiotherapy within 4 weeks or temozolomide within 14 days prior to registration or failure to recover from adverse events of either radiotherapy or temozolomide
* Patients may not be receiving any other investigational agents
* Severe, active comorbidity, defined as follows:

  * Any clinically significant cardiovascular disease including the following:

    * Unstable angina and/or congestive heart failure requiring hospitalization within the past 6 months
    * Transmural myocardial infarction or ventricular tachyarrhythmia within the past 6 months
    * Prolonged corrected QT interval (QTc) > 480 msec (Fridericia correction)
    * Ejection fraction less than institutional normal
    * Major conduction abnormality (unless a cardiac pacemaker is present)
  * Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration
  * Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at the time of registration
  * Acquired immune deficiency syndrome (AIDS) based upon current Centers for Disease Control and Prevention (CDC) definition; note, however, that human immunodeficiency virus (HIV) testing is not required for entry into this protocol
* Pregnancy or women of childbearing potential and men who are sexually active and not willing/able to use medically acceptable forms of contraception; breastfeeding should be discontinued if the mother is treated with dasatinib
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to dasatinib
* Patients who require concurrent treatment with any medications or substances that are potent inhibitors or inducers of cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP3A4) are ineligible
* Patients must not be taking hepatic enzyme inducing antiepileptic drugs (EIAEDs); if patients were previously on EIAEDs that have been discontinued, patients must have been off EIAEDs for >= 2 weeks prior to initiation of dasatinib
* Patients who require antacids should use short-acting, locally active agents (e.g., Maalox, Mylanta etc.); however, these agents should not be taken within either 2 hours before or 2 hours after the dasatinib dose
* Use of antithrombotic and/or antiplatelet agents (e.g., warfarin, heparin, low molecular weight heparin, aspirin, clopidogrel, ticlopidine, Aggrenox)
* Use of ibuprofen or non-steroidal anti-inflammatory drugs (NSAIDs)
* Patients with any condition (e.g., gastrointestinal tract disease resulting in an inability to take oral medication or a requirement for intravenous [IV] alimentation, prior surgical procedures affecting absorption, or active peptic ulcer disease) that impairs their ability to swallow and retain dasatinib tablets are excluded
* Prior treatment with stereotactic radiosurgery (including Gamma-Knife, Cyberknife, or other variants) or brachytherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2007-01-24 (Actual); Primary Completion 2011-03-09 (Actual); Study Completion 2018-09-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Lassman, Principal Investigator — NRG Oncology
Locations (188):
- United States (184):
  - Mobile Infirmary Medical Center, Mobile, Alabama
  - Arizona Oncology Services Foundation, Scottsdale, Arizona
  - The University of Arizona Medical Center-University Campus, Tucson, Arizona
  - Sutter Cancer Centers Radiation Oncology Services-Auburn, Auburn, California
  - Sutter Cancer Centers Radiation Oncology Services-Cameron Park, Cameron Park, California
  - Mercy San Juan Medical Center, Carmichael, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Glendale Adventist Medical Center, Glendale, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Sutter Cancer Centers Radiation Oncology Services-Roseville, Roseville, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Mercy General Hospital Radiation Oncology Center, Sacramento, California
  - Sutter Cancer Centers Radiation Oncology Services-Vacaville, Vacaville, California
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Boca Raton Regional Hospital, Boca Raton, Florida
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - University of Florida Health Science Center - Gainesville, Gainesville, Florida
  - Baptist MD Anderson Cancer Center, Jacksonville, Florida
  - Integrated Community Oncology Network-Southside Cancer Center, Jacksonville, Florida
  - University of Florida Health Science Center - Jacksonville, Jacksonville, Florida
  - Baptist Medical Center South, Jacksonville, Florida
  - Integrated Community Oncology Network-Florida Cancer Center Beaches, Jacksonville Beach, Florida
  - Jupiter Medical Center, Jupiter, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - 21st Century Oncology-Orange Park, Orange Park, Florida
  - 21st Century Oncology-Palatka, Palatka, Florida
  - Bay Medical Center, Panama City, Florida
  - Integrated Community Oncology Network-Flager Cancer Center, Saint Augustine, Florida
  - John B Amos Cancer Center, Columbus, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Saint John's Hospital, Springfield, Illinois
  - Saint Vincent Anderson Regional Hospital/Cancer Center, Anderson, Indiana
  - Franciscan Saint Francis Health-Beech Grove, Beech Grove, Indiana
  - IU Health Methodist Hospital, Indianapolis, Indiana
  - Reid Health, Richmond, Indiana
  - Menorah Medical Center, Overland Park, Kansas
  - Saint Luke's South Hospital, Overland Park, Kansas
  - Kansas City NCI Community Oncology Research Program, Prairie Village, Kansas
  - Shawnee Mission Medical Center-KCCC, Shawnee Mission, Kansas
  - The James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - Union Hospital of Cecil County, Elkton, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - Michigan Cancer Research Consortium NCORP, Ann Arbor, Michigan
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Beaumont Hospital-Dearborn, Dearborn, Michigan
  - Ascension Saint John Hospital, Detroit, Michigan
  - Green Bay Oncology - Escanaba, Escanaba, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Regional Medical Center-West Flint Campus, Flint, Michigan
  - Green Bay Oncology - Iron Mountain, Iron Mountain, Michigan
  - Allegiance Health, Jackson, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - Saint Mary's of Michigan, Saginaw, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview-Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Metro Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Singing River Hospital, Pascagoula, Mississippi
  - Cape Radiation Oncology, Cape Girardeau, Missouri
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Centerpoint Medical Center LLC, Independence, Missouri
  - Truman Medical Center, Kansas City, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Saint Joseph Health Center, Kansas City, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - Heartland Hematology and Oncology Associates Incorporated, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Liberty Radiation Oncology Center, Liberty, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Cancer Research for the Ozarks NCORP, Springfield, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Renown Regional Medical Center, Reno, Nevada
  - Cheshire Medical Center-Dartmouth-Hitchcock Keene, Keene, New Hampshire
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Virtua Memorial, Mount Holly, New Jersey
  - Sparta Cancer Treatment Center, Sparta, New Jersey
  - Virtua Voorhees, Voorhees Township, New Jersey
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Highland Hospital, Rochester, New York
  - University of Rochester, Rochester, New York
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Summa Akron City Hospital/Cooper Cancer Center, Akron, Ohio
  - Cleveland Clinic Akron General, Akron, Ohio
  - Summa Barberton Hospital, Barberton, Ohio
  - Aultman Health Foundation, Canton, Ohio
  - University of Cincinnati/Barrett Cancer Center, Cincinnati, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Health Center, Dayton, Ohio
  - Veteran Affairs Medical Center, Dayton, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - UH Seidman Cancer Center at Salem Regional Medical Center, Salem, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - University Pointe, West Chester, Ohio
  - Cancer Treatment Center, Wooster, Ohio
  - Greene Memorial Hospital, Xenia, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Salem Hospital, Salem, Oregon
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Delaware County Memorial Hospital, Drexel Hill, Pennsylvania
  - Northeast Radiation Oncology Center, Dunmore, Pennsylvania
  - Adams Cancer Center, Gettysburg, Pennsylvania
  - Cherry Tree Cancer Center, Hanover, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Upper Delaware Valley Cancer Center, Milford, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - WellSpan Health-York Hospital, York, Pennsylvania
  - AnMed Health Hospital, Anderson, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Eastside, Greenville, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Wellmont Holston Valley Hospital and Medical Center, Kingsport, Tennessee
  - Thompson Cancer Survival Center, Knoxville, Tennessee
  - Thompson Cancer Survival Center - West, Knoxville, Tennessee
  - Thompson Cancer Survival Center at Methodist, Oak Ridge, Tennessee
  - University of Texas Medical Branch, Galveston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Covenant Medical Center-Lakeside, Lubbock, Texas
  - American Fork Hospital / Huntsman Intermountain Cancer Center, American Fork, Utah
  - Sandra L Maxwell Cancer Center, Cedar City, Utah
  - Logan Regional Hospital, Logan, Utah
  - Cottonwood Hospital Medical Center, Murray, Utah
  - Intermountain Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center, Provo, Utah
  - Intermountain Health Care, Salt Lake City, Utah
  - Utah Cancer Specialists-Salt Lake City, Salt Lake City, Utah
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Dixie Medical Center Regional Cancer Center, St. George, Utah
  - University of Vermont Medical Center, Burlington, Vermont
  - University of Vermont College of Medicine, Burlington, Vermont
  - Norris Cotton Cancer Center-North, Saint Johnsbury, Vermont
  - Southwest VA Regional Cancer Center, Norton, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - Wheeling Hospital/Schiffler Cancer Center, Wheeling, West Virginia
  - Green Bay Oncology at Saint Vincent Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Green Bay Oncology Limited at Saint Mary's Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Bay Area Medical Center, Marinette, Wisconsin
  - Froedtert and the Medical College of Wisconsin, Milwaukee, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Green Bay Oncology - Oconto Falls, Oconto Falls, Wisconsin
  - Green Bay Oncology - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - ProHealth Waukesha Memorial Hospital, Waukesha, Wisconsin
- Canada (3):
  - London Regional Cancer Program, London, Ontario
  - CHU de Quebec-L'Hotel-Dieu de Quebec (HDQ), Québec, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
- King Faisal Specialist Hospital and Research Centre, Riyadh, Saudi Arabia

REFERENCES:
- [Derived] Lassman AB, Pugh SL, Gilbert MR, Aldape KD, Geinoz S, Beumer JH, Christner SM, Komaki R, DeAngelis LM, Gaur R, Youssef E, Wagner H, Won M, Mehta MP. Phase 2 trial of dasatinib in target-selected patients with recurrent glioblastoma (RTOG 0627). Neuro Oncol. 2015 Jul;17(7):992-8. doi: 10.1093/neuonc/nov011. Epub 2015 Mar 10. PMID 25758746

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Per protocol criteria, the study did not continue to Stage 2 and therefore no patients were accrued to this arm.
Groups:
- Stage 1: Dasatinib 200mg/Day: Patients receive oral 100mg dasatinib twice daily on days 1-28. Courses repeat every 28 days in the absence of disease progression and unacceptable toxicity
- Stage 1B: Dasatinib up to 400mg/Day; Stage 2: Dasatinib up to 400mg/Day: Patients begin with oral 100mg dasatinib twice daily on days 1-28. Courses repeat every 28 days in the absence of disease progression and unacceptable toxicity. Patients could escalate 50mg/day at each new cycle up to 400mg/day if they had not progressed to date and had not experienced dose-limiting toxicity.
Period: Overall Study
Arm/Group | Stage 1: Dasatinib 200mg/Day | Stage 1B: Dasatinib up to 400mg/Day | Stage 2: Dasatinib up to 400mg/Day
Started | 29 | 35 | 0
Completed | 21 | 29 | 0
Not Completed | 8 | 6 | 0
Not completed — Ineligible / No protocol treatment | 8 | 6 | 0

BASELINE CHARACTERISTICS:
Population: Eligible patients who started protocol treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Stage 1: Dasatinib 200mg/Day | Stage 1B: Dasatinib up to 400mg/Day | Stage 2: Dasatinib up to 400mg/Day | Total
Number analyzed (Participants) | 21 | 29 | 0 | 50
Age, Continuous [Median (Full Range); unit: years] | 51 [33 to 81] | 54 [26 to 75] |  | 54 [26 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 12 |  | 23
  Male | 10 | 17 |  | 27

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Achieving 6-month Progression-free Survival (6mPFS)
Description: This study utilized a two-stage phase II design (Stage 1B and 2). The primary endpoint of 6-month progression-free survival (6mPFS) would be assessed based on the patients combined from 1B and 2 if the study continued to Stage 2. Null hypothesis = 11%; alternative hypothesis = 25%. Simon's minmax 2-stage design was used with type I and type II error both set at 10%. If the first stage met its criteria (see secondary outcome measure), then accrual would continue, otherwise there would be no further accrual and the alternative hypothesis would be rejected. Following Stage 2 accrual completion and 6 months of follow-up, if 9 or more patients were alive without progression by 6 months, the null hypothesis would be rejected in favor of the alternative.
Time Frame: Registration to 6 months
Population: Eligible patients who started protocol treatment.
Measure: Number; unit: participants
Groups:
- Stage 2:: Patients begin with oral 100mg dasatinib twice daily on days 1-28. Courses repeat every 28 days in the absence of disease progression and unacceptable toxicity. Patients could escalate 50mg/day at each new cycle up to 400mg/day if they had not progressed to date and had not experienced dose-limiting toxicity
Arm/Group | Stage 1: Dasatinib 200mg/Day | Stage 1B: Dasatinib up to 400mg/Day | Stage 2:
Number analyzed (Participants) | 21 | 29 | 0
participants | 1 | 2 |

2. Secondary Outcome: Number of Patients Achieving Objective Response (Partial or Complete Response) OR 6-month Progression-free Survival (6mPFS)
Description: Study design and efficacy determination uses the hybrid endpoint of 6mPFS or complete/partial response of any duration prior to or at 6 months. Null hypothesis = 11%; alternative hypothesis = 25%. Simon's minmax 2-stage design was used with type I and type II error both set at 10%. Stage 1 and 1B: If 2 or fewer patients were alive and progression-free at 6 months or achieved complete/partial response, then there would be no further accrual and the alternative hypothesis would be rejected. Otherwise accrual would continue to a total of 50 analyzable patients to address the primary endpoint. Complete Response: Complete disappearance of all enhancing tumor on consecutive CT or MRI scans at least 1 month apart; off corticosteroids; neurologically stable/improved. Partial Response: ≥ 50% decrease in size of enhancing tumor on consecutive CT or MRI scans at least 1 month apart; corticosteroids stable/reduced; neurologically stable/improved.
Time Frame: Registration to 6 months
Population: Eligible patients who started protocol treatment.
Measure: Number; unit: participants
Arm/Group | Stage 1: Dasatinib 200mg/Day | Stage 1B: Dasatinib up to 400mg/Day
Number analyzed (Participants) | 21 | 29
participants | 1 | 2

3. Secondary Outcome: Overall Survival
Description: Survival time is defined as time from randomization to date of death from any cause and is estimated by the Kaplan-Meier method. Patients last known to be alive are censored at the date of last contact. The study is not designed for a comparison of the treatment arms to each other.
Time Frame: Analysis occurs after all patients have been on study for at least 6 months. (Patients are followed from registration to death or study termination whichever occurs first.)
Population: Survival time is defined as time from randomization to date of death from any cause and is estimated by the Kaplan-Meier method. Patients last known to be alive are censored at the date of last contact. This analysis was planned to occur when all patients had been potentially followed for at least 6 months. Arms are not compared.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Stage 1: Dasatinib 200mg/Day | Stage 1B: Dasatinib up to 400mg/Day
Number analyzed (Participants) | 21 | 29
months | 6.5 [3.5 to 9.5] | 8.9 [5.0 to 11.3]

4. Secondary Outcome: Treatment Response Rates at Six Months
Description: Best response is assessed using standard criteria for patients with malignant gliomas (Macdonald 1990) as reported by the site. Complete response (CR): Complete disappearance of all enhancing tumor on consecutive CT or MRI scans at least 1 month apart; off corticosteroids; neurologically stable/improved. Partial response (PR): ≥ 50% decrease in size of enhancing tumor on consecutive CT or MRI scans at least 1 month apart; corticosteroids stable/reduced; neurologically stable/improved. Stable disease (SD): Does not qualify for CR, PR, or PD. Progressive disease (PD): ≥ 25% increase in the size of enhancing tumor or any new tumor; neurologically worse; steroids stable/increased. The best tumor response is defined as the best radiographic response for patients evaluable for radiographic response prior to progression, up to six months. The study is not designed for a comparison of the treatment arms to each other.
Time Frame: From registration to 6 months
Population: Eligible patients who started study treatment
Measure: Number; unit: percentage of participants
Arm/Group | Stage 1: Dasatinib 200mg/Day | Stage 1B: Dasatinib up to 400mg/Day
Number analyzed (Participants) | 21 | 29
percentage of participants
  CR or PR | 0.0 | 0.0
  Stable | 19.0 | 27.6
  Progression | 76.2 | 69.0
  No scan done and no clinical progression reported | 4.8 | 3.4

5. Secondary Outcome: Progression-free Survival
Description: Progression-free survival time is measured from randomization to the date of first progression or death, else the last follow-up date on which the patient was reported alive, and is estimated by the Kaplan-Meier method. Progression is defined as ≥ 25% increase in the size of enhancing tumor or any new tumor, neurologically worse, or steroids stable/increased. The study is not designed for a comparison of the treatment arms to each other.
Time Frame: as for outcome 3
Population: Eligible patients who started study treatment
Measure: Mean (95% Confidence Interval); unit: months
Arm/Group | Stage 1: Dasatinib 200mg/Day | Stage 1B: Dasatinib up to 400mg/Day
Number analyzed (Participants) | 21 | 29
months | 1.7 [1.0 to 2.0] | 1.8 [1.2 to 2.0]

6. Secondary Outcome: Rate of Adverse Events
Description: The rate of patients' worst overall grade of adverse event is reported. Adverse events are graded using CTCAE v3.0. Grade refers to the severity of the AE. The CTCAE v3.0 assigns Grades 1 through 5 with unique clinical descriptions of severity for each AE based on this general guideline: Grade 1 Mild AE, Grade 2 Moderate AE, Grade 3 Severe AE, Grade 4 Life-threatening or disabling AE, Grade 5 Death related to AE. The study is not designed for a comparison of the treatment arms to each other.
Time Frame: as for outcome 3
Population: Eligible patients who started protocol treatment
Measure: Number; unit: percentage of participants
Arm/Group | Stage 1: Dasatinib 200mg/Day | Stage 1B: Dasatinib up to 400mg/Day
Number analyzed (Participants) | 21 | 29
percentage of participants
  Grade 1 | 0.0 | 10.3
  Grade 2 | 14.3 | 17.2
  Grade 3 | 57.1 | 44.8
  Grade 4 | 14.3 | 3.4
  Grade 5 | 14.3 | 17.2

7. Secondary Outcome: Correlation of Molecular Markers and Tumor Response
Description: The following markers were examined: p-SRC, PDGFR, EPHA2, c-KIT. Patients were categorized based on the number of positive molecular markers they had: 2 vs. 3 and 4. Correlation of marker category and best tumor response was tested using Fisher's exact test. The best tumor response is defined as the best radiographic response for patients evaluable for radiographic response prior to progression up to six months. Patients are combined from the two treatment arms.
Time Frame: From registration to 6 months
Population: Eligible patients who started study treatment and whose response was assessed
Measure: Count of Participants; unit: Participants
Groups:
- Stable Disease: Patients with best response of "stable disease" by six months. Stable disease (SD): Does not qualify for CR, PR, or PD. Progressive disease (PD): ≥ 25% increase in the size of enhancing tumor or any new tumor, neurologically worse, or steroids stable/increased.
- Progressive Disease: Patients with best tumor response of "progressive disease" by six months. Progressive disease (PD): ≥ 25% increase in the size of enhancing tumor or any new tumor, neurologically worse, or steroids stable/increased.
Arm/Group | Stable Disease | Progressive Disease
Number analyzed (Participants) | 12 | 36
Participants
  2 postivie molecular markers | 4 | 13
  3 or 4 positive molecular markers | 8 | 23
Statistical Analysis 1: Comparison: Stable Disease vs Progressive Disease; Test type: Superiority; p = 0.99, Fisher Exact; 2-sided test

8. Secondary Outcome: Correlation of Pharmacokinetic Data With Dosing, Toxicity, and Efficacy
Description: Sufficient pharmacokinetic data was not obtained.
Time Frame: as for outcome 3
Arm/Group | Stage 1: Dasatinib 200mg/Day | Stage 1B: Dasatinib up to 400mg/Day
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: Subjects experiencing more than one of a given serious adverse event (SAE) are counted only once for that SAE. The same methodology was applied for non-SAE adverse events (AE).
Groups:
- Stage 1: Dasatinib 200mg/Day: Patients receive oral 100mg dasatinib twice daily on days 1-28. Courses repeat every 28 days in the absence of disease progression and unacceptable toxicity
  dasatinib: Given orally
- Stage 1B: Dasatinib up to 400mg/Day: Patients begin with oral 100mg dasatinib twice daily on days 1-28. Courses repeat every 28 days in the absence of disease progression and unacceptable toxicity. Patients could escalate 50mg/day at each new cycle up to 400mg/day if they had not progressed to date and had not experienced dose-limiting toxicity.
  dasatinib: Given orally
Arm/Group | Stage 1: Dasatinib 200mg/Day | Stage 1B: Dasatinib up to 400mg/Day
Serious Adverse Events (participants affected / at risk) | 8/21 | 14/29
Other Adverse Events (participants affected / at risk) | 21/21 | 23/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stage 1: Dasatinib 200mg/Day (N=21) | Stage 1B: Dasatinib up to 400mg/Day (N=29)
Hemoglobin (Blood and lymphatic system disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 0
Anal haemorrhage (Gastrointestinal disorders) | 1 | 0
Colitis NOS (Gastrointestinal disorders) | 1 | 0
Diarrhoea NOS (Gastrointestinal disorders) | 1 | 0
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1
Vomiting NOS (Gastrointestinal disorders) | 0 | 1
Chest pain (General disorders) | 0 | 1
Constitutional Symptoms - Other: (General disorders) | 1 | 0
Disease progression NOS (General disorders) | 1 | 4
Fatigue (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 1
Rigors (General disorders) | 0 | 1
Infection - Other: (Infections and infestations) | 0 | 1
Lymphopenia (Investigations) | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 0 | 2
Dehydration (Metabolism and nutrition disorders) | 2 | 1
Hyperglycaemia NOS (Metabolism and nutrition disorders) | 1 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycemia NOS (Metabolism and nutrition disorders) | 1 | 0
Muscle weakness, generalized or specific area (not due to neuropathy): Extremity-lower (Musculoskeletal and connective tissue disorders) | 0 | 1
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 1
Convulsions NOS (Nervous system disorders) | 2 | 3
Depressed level of consciousness (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 2
Peripheral motor neuropathy (Nervous system disorders) | 0 | 2
Syncope (Nervous system disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 2
Renal failure NOS (Renal and urinary disorders) | 1 | 0
Dermatitis exfoliative NOS (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatology/skin - Other: (Skin and subcutaneous tissue disorders) | 0 | 1
Hematoma (Vascular disorders) | 1 | 0
Hypotension NOS (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stage 1: Dasatinib 200mg/Day (N=21) | Stage 1B: Dasatinib up to 400mg/Day (N=29)
Blood/bone marrow - Other: (Blood and lymphatic system disorders) | 2 | 0
Hemoglobin (Blood and lymphatic system disorders) | 13 | 12
Cardiac General - Other: (Cardiac disorders) | 2 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 3 | 0
Ventricular arrhythmia NOS (Cardiac disorders) | 0 | 1
Auditory/ear - Other: (Ear and labyrinth disorders) | 2 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0
Cushingoid (Endocrine disorders) | 2 | 0
Dry eye NOS (Eye disorders) | 1 | 0
Extraocular muscle disorder (Eye disorders) | 1 | 1
Ocular/visual - Other: (Eye disorders) | 1 | 1
Vision blurred (Eye disorders) | 1 | 1
Abdominal pain NOS (Gastrointestinal disorders) | 2 | 1
Anal haemorrhage (Gastrointestinal disorders) | 1 | 0
Colitis NOS (Gastrointestinal disorders) | 0 | 1
Colonic perforation (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 6 | 3
Diarrhoea NOS (Gastrointestinal disorders) | 13 | 7
Dry mouth (Gastrointestinal disorders) | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 2 | 2
Faecal incontinence (Gastrointestinal disorders) | 0 | 1
Gastrointestinal - Other: (Gastrointestinal disorders) | 0 | 1
Hemorrhoids (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 7 | 11
Oral pain (Gastrointestinal disorders) | 0 | 1
Proctalgia (Gastrointestinal disorders) | 1 | 0
Proctitis NOS (Gastrointestinal disorders) | 1 | 0
Rectal hemorrhage (Gastrointestinal disorders) | 1 | 0
Stomach discomfort (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1
Vomiting NOS (Gastrointestinal disorders) | 4 | 8
Constitutional Symptoms - Other: (General disorders) | 1 | 0
Death NOS (General disorders) | 1 | 0
Disease progression NOS (General disorders) | 1 | 0
Edema: head and neck: (General disorders) | 3 | 4
Edema: limb: (General disorders) | 7 | 4
Fatigue (General disorders) | 14 | 20
Gait abnormal NOS (General disorders) | 3 | 2
Pain - Other: (General disorders) | 1 | 0
Pain NOS (General disorders) | 1 | 0
Pyrexia (General disorders) | 3 | 2
Rigors (General disorders) | 0 | 1
Autoimmune disorder NOS (Immune system disorders) | 1 | 0
Abdominal infection (Infections and infestations) | 0 | 1
Eye infection NOS (Infections and infestations) | 1 | 1
Gingival infection (Infections and infestations) | 0 | 1
Infection - Other: (Infections and infestations) | 1 | 0
Infection with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L): Oral cavity-gums (gingivitis) (Infections and infestations) | 1 | 0
Infection with normal ANC or Grade 1 or 2 neutrophils: Colon (Infections and infestations) | 1 | 0
Infection with unknown ANC: Colon (Infections and infestations) | 1 | 0
Opportunisitic infection (Infections and infestations) | 1 | 1
Respiratory tract infection NOS (Infections and infestations) | 0 | 1
Urinary tract infection NOS (Infections and infestations) | 1 | 1
Burn: (Injury, poisoning and procedural complications) | 1 | 0
Culture wound negative (Injury, poisoning and procedural complications) | 0 | 1
Ecchymosis (Injury, poisoning and procedural complications) | 3 | 1
Alanine aminotransferase increased (Investigations) | 11 | 8
Aspartate aminotransferase increased (Investigations) | 6 | 6
Blood alkaline phosphatase increased (Investigations) | 4 | 1
Blood bilirubin increased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 1 | 1
Hypercholesterolaemia (Investigations) | 1 | 0
Leukopenia NOS (Investigations) | 7 | 6
Lymphopenia (Investigations) | 9 | 5
Metabolic/laboratory - Other: (Investigations) | 8 | 2
Neutrophil count (Investigations) | 3 | 3
Platelet count decreased (Investigations) | 6 | 7
Troponin I increased (Investigations) | 1 | 0
Weight decreased (Investigations) | 4 | 3
Weight increased (Investigations) | 2 | 0
Anorexia (Metabolism and nutrition disorders) | 7 | 5
Dehydration (Metabolism and nutrition disorders) | 3 | 1
Hyperglycaemia NOS (Metabolism and nutrition disorders) | 14 | 10
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypermagnesaemia (Metabolism and nutrition disorders) | 1 | 2
Hypernatremia (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 8 | 6
Hypocalcemia (Metabolism and nutrition disorders) | 10 | 10
Hypoglycemia NOS (Metabolism and nutrition disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 4 | 8
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 3 | 4
Hypophosphataemia (Metabolism and nutrition disorders) | 4 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint disorder NOS (Musculoskeletal and connective tissue disorders) | 1 | 1
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle weakness NOS (Musculoskeletal and connective tissue disorders) | 3 | 6
Muscle weakness, generalized or specific area (not due to neuropathy): Extremity-lower (Musculoskeletal and connective tissue disorders) | 5 | 1
Muscle weakness, generalized or specific area (not due to neuropathy): Extremity-upper (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle weakness, generalized or specific area (not due to neuropathy): Left-sided (Musculoskeletal and connective tissue disorders) | 1 | 1
Musculoskeletal/soft tissue - Other: (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 4
Ataxia (Nervous system disorders) | 1 | 1
Cognitive disorder (Nervous system disorders) | 1 | 1
Convulsions NOS (Nervous system disorders) | 1 | 7
Depressed level of consciousness (Nervous system disorders) | 1 | 3
Dizziness (Nervous system disorders) | 1 | 2
Dysgeusia (Nervous system disorders) | 2 | 1
Facial nerve disorder NOS (Nervous system disorders) | 2 | 0
Headache (Nervous system disorders) | 8 | 10
Hyperreflexia (Nervous system disorders) | 2 | 2
Hypoglossal nerve disorder NOS (Nervous system disorders) | 0 | 1
Memory impairment (Nervous system disorders) | 2 | 4
Neuralgia NOS (Nervous system disorders) | 1 | 0
Neuropathy: cranial: CN VIII Hearing and balance (Nervous system disorders) | 1 | 0
Peripheral motor neuropathy (Nervous system disorders) | 1 | 2
Peripheral sensory neuropathy (Nervous system disorders) | 3 | 4
Speech disorder (Nervous system disorders) | 5 | 4
Tremor (Nervous system disorders) | 2 | 0
VIth nerve disorder (Nervous system disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 3 | 4
Confusional state (Psychiatric disorders) | 2 | 1
Depression (Psychiatric disorders) | 3 | 3
Insomnia (Psychiatric disorders) | 4 | 6
Pollakiuria (Renal and urinary disorders) | 2 | 5
Proteinuria (Renal and urinary disorders) | 2 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 2
Urogenital hemorrhage (Renal and urinary disorders) | 1 | 1
Muscle weakness, generalized or specific area (not due to neuropathy): Pelvic (Reproductive system and breast disorders) | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal cavity/paranasal sinus reactions: (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pulmonary/upper respiratory - Other: (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinitis allergic NOS (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acne NOS (Skin and subcutaneous tissue disorders) | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 5 | 2
Dermatitis exfoliative NOS (Skin and subcutaneous tissue disorders) | 8 | 6
Dermatology/skin - Other: (Skin and subcutaneous tissue disorders) | 2 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 2
Pain of skin (Skin and subcutaneous tissue disorders) | 2 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 1
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 2 | 0
Flushing (Vascular disorders) | 3 | 0
Hematoma (Vascular disorders) | 1 | 0
Hemorrhage/bleeding - Other: (Vascular disorders) | 2 | 0
Hot flushes NOS (Vascular disorders) | 3 | 1
Hypertension NOS (Vascular disorders) | 1 | 1
Hypotension NOS (Vascular disorders) | 1 | 2
Lymphoedema NOS (Vascular disorders) | 1 | 0
Thrombosis (Vascular disorders) | 2 | 0
Vascular - Other: (Vascular disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
Designed as a 2-stage study. The protocol was amended after Stage 1 to add Stage 1B allowing intra-patient escalation. Per protocol criteria, the study did not continue to Stage 2.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less